CLINICAL TRIAL: NCT02318004
Title: Study Protocol for Evaluation of EarlySense Home Care Tele-monitoring Device - A Contact-Free System for Measuring Heart Rate, Respiratory Rate and Motion For Early Detection of Deterioration For Cardiac Patients at Home
Brief Title: Evaluation of EarlySense Home Care Tele-monitoring Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: EarlySense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-14-0987-RK-CTIL
Record Dates: First submitted 2014-12-07; First posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Myocardial Infarction; Cardiac Surgery
Keywords: telemonitoring
MeSH Terms: conditions — Myocardial Infarction | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home monitoring (Experimental): Home monitoring via the EarlySense non-invasive nocturnal monitoring system. Movement, heart rate and respiratory rates will be monitored while subject is in his bed. The trends of monitored values will be daily reported to a central repository. No intervention will be attempted and care will be coordinated by the family physician and treating cardiologist as usual.
  Interventions: Other: Home Monitoring

INTERVENTIONS:
Other: Home Monitoring — Non invasive nocturnal monitoring of heart and respiratory rate and subjects movement out of bed.

SUMMARY:
The aims of the present study are to evaluate the information obtained by the EarlySenese monitoring system and examine correlation of the obtained data and clinical events.

DETAILED DESCRIPTION:
The EarlySense Home Care System developed by EarlySense, Ltd., is a contact-less tele-monitoring system. The system is intended for continuous monitoring of patients' respiration rate, heart rate and patient's motion.

The system, which monitors the patient while in bed, consists of a piezoelectric sensor that produces an electrical signal in response to physiological stimulation, and a microprocessor control unit that analyzes the recorded signal and identifies respiratory and heart rates and patient motion, while patient is in bed,. In addition, the system indicates patient's in or out of bed status. The system also provides alerts if either of the physiological parameters cross predefined threshold settings (e.g., high/ low heart rate or respiratory rate, or motion or time in bed).

The system saves patient's parameters and then flags the patients, as those to have changes in their vital signs and motion, or those that do not have noteworthy changes during recent hours of monitoring. Flagging of the patients are based on changes detected in patients' baseline vital signs (heart and respiratory rates and patterns) and well as recognition of changes in patients motion and in and out of bed status in comparison to set thresholds.

The aim of this study is to evaluate relevance of the information (vital sign trends, alerts and flags) as provided by the EarlySense Home Care Tele-monitoring system to medical staff in Sheba Medical Center's Heart Rehabilitation Institute (Shelev) in order proactively monitor patients at home. The correlation between the EarlySense system alerts and flags to patient deterioration and hospital readmission will be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who resided in Shelev following a cardiac event (cardiac surgery, myocardial infarction, pacemaker implantation or other cardiac interventions )
2. Age ≥ 21 years
3. Any patient hosted in Shelev with geographically resident within 50 Km from Sheba Medical Center
4. Patients agrees to sign the consent form and able to comply with study protocol.
5. Sleeps on a mattress

Exclusion Criteria:

1. Planned readmission within 30 days of discharge from hospital
2. Discharge to hospice care.
3. Patients with cognitive disabilities
4. Patient's major treating hospital is not the Sheba Medical Center

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Diagnositic Utility | 30 days following enrollment
  Positive percent agreement between the EarlySense device and clinical events as adjudicated by health-care personal

SECONDARY OUTCOMES:
System Acceptance | 30 days following enrollment
  Assess the acceptability of the EarlySense Home care device by clinicians and by patients and their families in their own home as determined by a provided questioner.

CONTACTS AND LOCATIONS:
Locations (1):
- SheLev, Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Zimlichman E, Szyper-Kravitz M, Shinar Z, Klap T, Levkovich S, Unterman A, Rozenblum R, Rothschild JM, Amital H, Shoenfeld Y. Early recognition of acutely deteriorating patients in non-intensive care units: assessment of an innovative monitoring technology. J Hosp Med. 2012 Oct;7(8):628-33. doi: 10.1002/jhm.1963. Epub 2012 Aug 3. PMID 22865462
- [Background] Zimlichman E, Shinar Z, Rozenblum R, Levkovich S, Skiano S, Szyper-Kravitz M, Altman A, Amital H, Shoenfeld Y. Using continuous motion monitoring technology to determine patient's risk for development of pressure ulcers. J Patient Saf. 2011 Dec;7(4):181-4. doi: 10.1097/PTS.0b013e318230e6ef. PMID 21926639